CLINICAL TRIAL: NCT01569763
Title: Minerva Pivotal Study
Brief Title: Minerva Pivotal Study to Evaluate Safety and Efficacy of the Aurora Endometrial Ablation System Compared to Hysteroscopic Rollerball Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minerva Surgical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIP0005
Record Dates: First submitted 2012-03-30; First posted 2012-04-03 (Estimated); Results first posted 2016-05-05 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-03

CONDITIONS: Menorrhagia
Keywords: endometrial ablation
MeSH Terms: conditions — Menorrhagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hysteroscopic rollerball resection/ablation (Active Comparator)
  Interventions: Device: Rollerball Ablation/Resection
- Aurora Endometrial Ablation (Experimental)
  Interventions: Device: Aurora Endometrial Ablation

INTERVENTIONS:
Device: Aurora Endometrial Ablation — Endometrial Ablation using the Aurora Endometrial Ablation system
  Arms: Aurora Endometrial Ablation
Device: Rollerball Ablation/Resection — Hysteroscopic rollerball resection/ablation
  Arms: hysteroscopic rollerball resection/ablation

SUMMARY:
The primary objective of this study is to evaluate the safety and effectiveness of the Aurora Endometrial Ablation System as compared to hysteroscopic rollerball endometrial ablation in reducing menstrual blood loss at 12 months post-treatment.

DETAILED DESCRIPTION:
Menorrhagia is defined as menstrual bleeding in the ovulatory woman exceeding 80 ml per month. Approximately 20-25% of healthy premenopausal women have abnormal uterine bleeding. Menorrhagia can have a negative impact on a woman's lifestyle and self-perception, often leading her to seek definitive treatment. Pharmacologic treatment for menorrhagia is not always successful, and dilatation and curettage typically provides relief for only a few menstrual cycles. Traditionally hysterectomy has been the definitive treatment for menorrhagia. This clinical study evaluates the safety and effectiveness of the Aurora Endometrial Ablation System to provide a therapeutic treatment for menorrhagia due to benign causes by ablating the endometrial lining of the uterus in pre-menopausal women for whom childbearing is complete. Subjects who are randomized to the control group will receive hysteroscopic rollerball/resection ablation. Subjects randomized to the test arm will be treated with the Aurora Endometrial Ablation System.

ELIGIBILITY:
Inclusion Criteria:

* Refractory menorrhagia with no definable organic cause
* Female subject from (and including) age 25 to 50 years
* Uterine sound measurement of no greater than10.0cm (external os to internal fundus) and a minimum uterine cavity length of 4.0cm
* A minimum menstrual blood loss of ≥ 160 ml for two baseline cycles within three months prior to treatment as measured by alkaline hematin extraction; OR,

  * A minimum menstrual blood loss of ≥ 160 ml for one baseline cycle for women who either
  * had at least 3 prior months documented failed medical therapy; or
  * had a contraindication to medical therapy
* Premenopausal at enrollment as determined by FSH measurement ≤ 40 IU/L
* Not pregnant and no desire to conceive at any time
* Subject agrees to use a reliable form of contraception up to the 12-month follow-up visit. If a hormonal birth control method is used for contraception, the subject must have been on said method for ≥ 3 months prior to enrollment and agrees to remain on the same hormonal regimen through the initial 12-month follow-up
* Able to provide written informed consent using a form that has been approved by the reviewing IRB/EC
* Subject agrees to follow-up exams and data collection requirements
* Subject who is literate or demonstrates an understanding on how to collect menstrual blood loss products for the alkaline hematin method of analysis

Exclusion Criteria:

* Pregnancy or subject with a desire to conceive
* Endometrial hyperplasia as confirmed by histology
* Presence of active endometritis
* Active pelvic inflammatory disease
* Active sexually transmitted disease (STD)
* Presence of bacteremia, sepsis, or other active systemic infection
* Active infection of the genitals, vagina, cervix, uterus or urinary tract at the time of the procedure
* Known/suspected abdominal pelvic or gynecological malignancy within the past 5 years
* Known clotting defects or bleeding disorders
* Untreated/unevaluated cervical dysplasia, except CIN I
* Prior uterine surgery (except low segment cesarean section) that interrupts the integrity of the uterine wall (e.g., transmural myomectomy or classical cesarean section)
* Previous endometrial ablation procedure
* Presence of an implantable (intrauterine) contraceptive device (e.g. Essure™ or Adiana™)
* Currently on medications that could thin the myometrial muscle, such as long-term steroid use (except inhaler or nasal therapy for asthma)
* Currently on anticoagulants
* Abnormal or obstructed cavity as confirmed by hysteroscopy, SIS or vaginal ultrasound
* Presence of an intrauterine device (IUD) which the Subject is unwilling to have removed at the time of the operative visit
* Subject currently on hormonal birth control therapy (including the Mirena device) for <3 months prior to enrollment
* Subject who is unwilling to use birth control post-ablation whether non-hormonal birth control or the same hormonal birth control therapy as before the procedure
* Subject who is within 6-weeks post partum
* Any subject who is currently participating or considers future participation in a research study of an investigational drug or device during the course of this investigational study
* Any general health condition which, in the opinion of the Investigator, could represent an increased risk for the subject

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 153 (Actual)
Dates: Start 2012-03; Primary Completion 2015-01 (Actual); Study Completion 2018-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Skalnyi, MD, Study Director — Minerva Surgical, Inc.
Locations (13):
- United States (8):
  - New Horizons Women's Care, Chandler, Arizona
  - Women's Health Research, Phoenix, Arizona
  - Basinski, LLC, Newburgh, Indiana
  - Cypress Medical Research Center, LLC, Wichita, Kansas
  - Minnesota Gynecology and Surgery, Edina, Minnesota
  - Mercy Clinic Minimally Invasive Gynecology, St Louis, Missouri
  - Tennessee Women's Care PC, Nashville, Tennessee
  - Baylor Research Institute, Fort Worth, Texas
- Canada (4):
  - McMaster University/Hamilton Health Sciences, Hamilton, Ontario
  - La Cite Medicale, Québec, Quebec
  - Hôpital LaSalle, Ville Lassalle, Quebec
  - Regina Qu'Appelle Health Region, Regina, Saskatchewan
- Hospital Universitario, UANL, Monterrey, Nuevo León, Mexico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled in the clinical trial at 13 Investigational Sites in the U.S., Canada, and Mexico between March 2012 until November 2013.
Pre-assignment Details: A total of 153 subjects were enrolled and randomized 2:1 to the Minerva (Aurora) Test Group (n=102) or the Rollerball Control Group (n=51). As part of the randomization process, subjects were stratified by age, though there was no attempt to enroll an equal number into the < 40 and > 40 age groups. All 153 subjects were successfully treated.
Period: Overall Study
Arm/Group | Aurora Endometrial Ablation | Hysteroscopic Rollerball Resection/Ablation
Started | 102 | 51
Treated | 102 | 51
Completed | 99 (Completed 12 Months of Follow-up) | 44 (Completed 12 Months of Follow-up)
Not Completed | 3 | 7
Not completed — Lack of Efficacy | 2 | 7
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: Enrolled Subjects
Groups:
- Aurora Endometrial Ablation: Aurora Endometrial Ablation: Endometrial Ablation using the Minerva Endometrial Ablation system
- Total: Total of all reporting groups
Arm/Group | Aurora Endometrial Ablation | Hysteroscopic Rollerball Resection/Ablation | Total
Number analyzed (Participants) | 102 | 51 | 153
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (4.2) | 42.5 (4.7) | 42.5 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 51 | 153
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 54 | 26 | 80
  United States | 20 | 12 | 32
  Mexico | 28 | 13 | 41
Alkaline Hematin Value at Baseline [Mean (Standard Deviation); unit: Menstrual Blood Loss (ml)] — Alkaline hematin methodology is a quantitative laboratory method used to evaluate the volume of menstrual blood loss, by collecting used sanitary products (tampons and pads) and extracting alkaline hematin from the hemoglobin from menstrual fluids.
  Menstrual Blood Loss (ml) | 310.2 (169.0) | 301.8 (176.1) | 307.4 (170.9)

OUTCOME MEASURES:

1. Primary Outcome: Reduction of Menstrual Bleeding to Normal or Below Normal at 12 Months
Description: Clinical success was defined as a reduction in menstrual bleeding volume to ≤ 80 ml as measured by the alkaline hematin method (AH). Clinical success was not achieved if: (1) at one year post-treatment menstrual blood loss is greater than 80ml, as measured by AH; (2) an acute failure occurred (e.g., aborted procedure, etc.); or (3) the subject required additional therapy to control menorrhagia.
Time Frame: 12 months
Population: All Randomized subjects in whom treatment was attempted
Measure: Number; unit: participants
Arm/Group | Aurora Endometrial Ablation | Hysteroscopic Rollerball Resection/Ablation
Number analyzed (Participants) | 102 | 51
participants | 95 | 41

2. Secondary Outcome: Procedure Time
Description: Procedure time is defined as the time from device insertion to time of device removal.
Time Frame: < 1 hour
Population: Subjects completing treatment
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Aurora Endometrial Ablation | Hysteroscopic Rollerball Resection/Ablation
Number analyzed (Participants) | 102 | 51
Minutes | 3.1 (0.5) | 17.2 (6.7)

3. Post Hoc Outcome: Subjects With Amenorrhea at 12 Months
Description: Amenorrhea at 12 Months- Number of Subjects experiencing no menstrual bleeding
Time Frame: 12 Months
Population: Randomized subjects
Measure: Number; unit: participants
Arm/Group | Aurora Endometrial Ablation | Hysteroscopic Rollerball Resection/Ablation
Number analyzed (Participants) | 102 | 51
participants | 73 | 25

ADVERSE EVENTS:
Time Frame: 1 year
Description: All Serious Adverse Events observed during the clinical study, regardless of relationship to the study device or procedure are reported below. All non-Serious Adverse Events considered possibly, probably or highly probably related to the device or procedure are reported below.
Arm/Group | Aurora Endometrial Ablation | Hysteroscopic Rollerball Resection/Ablation
Serious Adverse Events (participants affected / at risk) | 5/102 | 3/51
Other Adverse Events (participants affected / at risk) | 14/102 | 10/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aurora Endometrial Ablation (N=102) | Hysteroscopic Rollerball Resection/Ablation (N=51)
Bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Endometritis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic Inflammatory Disease (PID) (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Anesthesia Related (Surgical and medical procedures) | 1 (1) | 0 (0)
Thyroid Nodule (Endocrine disorders) | 1 (1) | 0 (0)
Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Continued Heavy Menstrual Bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aurora Endometrial Ablation (N=102) | Hysteroscopic Rollerball Resection/Ablation (N=51)
Skin Rash and/or Itching or Burning Sensation (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Bleeding or spotting (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Nausea and/or Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Backache (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fever (Surgical and medical procedures) | 1 (1) | 0 (0)
Abdominal Pain and/or Bloating (Gastrointestinal disorders) | 3 (3) | 2 (2)
Pelvic Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal discharge, unpleasant smell, burning, abnormal sensation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Weaknes, Fatigue, Sleepiness, Lack of concentration, Dizziness (General disorders) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Endometritis or Endomyometritis (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Pelvic Inflammatory Disease (PID) (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Hematometra (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dysmenorrhea (Reproductive system and breast disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator has the right to publish their research for non-profit and academic purposes, provided the 1st publication of results shall be in conjunction with results from all centers in this Study. If Investigator desires to publish/present data obtained by Investigator, following completion of the Study at all sites, Investigator may do so, provided a copy of proposed publication/presentation is received by Company for review/comment at least 15 days in advance of submission for publication.